CLINICAL TRIAL: NCT00142506
Title: This Protocol is a Randomized Prospective Study Comparing Prophylactic and on Demand Sildenafil Citrate Usage Administered During and After Radiotherapy With or Without Hormone Therapy Versus Radiotherapy With or Without Hormone Therapy Alone for the Preservation of Erectile Function After Therapy for Potent Patients With Clinically Localized Prostate Cancer
Brief Title: Study of Sildenafil Citrate During and After Radiotherapy/Hormone Therapy for Erectile Function Versus Radiotherapy/Hormone Therapy for Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Beth Israel Medical Center (Other); St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-007
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer; Erectile Dysfunction
Keywords: Prostate Cancer; Cancer of the Prostate; Prostate Neoplasms; Prostatic Cancer; Viagra; 05-007
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): radiotherapy with hormones, questionaire assessments
  Interventions: Drug: sildenafil citrate and questionaires
- 2 (Placebo Comparator): radiotherapy without hormones, questionaire assessments
  Interventions: Drug: placebo tablets and questionaires

INTERVENTIONS:
Drug: sildenafil citrate and questionaires — Hormone therapy patients will be instructed to begin the study drug simultaneously or within 1 month of start of hormone therapy. These patients will then continue to take the study drug for approximately 6 months following start of radiotherapy.In addition, during prophylactic phase (drug and placebo prophylactic arms) patients will have the opportunity to utilize oral 50 mg. tablets of Sildenafil Citrate in an on demand open label, flexible dose fashion. Hormone patients will be offered on demand Sildenafil for approximately 15-21 months.
  Hormone therapy patients will complete assessments at baseline (within 4 weeks of start of study treatment) each month (only IIEF and QOL) before start of radiotherapy, at start of radiotherapy and at months 3, 6, 9, 12 18 and 24 from start of radiotherapy. Testosterone assessments will take place at baseline, and months 12 and 24.
  Arms: 1
Drug: placebo tablets and questionaires — Non-hormone therapy patients will be instructed to begin the study drug 3 days prior to start of radiotherapy. Patients beginning study drug anytime between 3 days before start of radiotherapy and 2 weeks after the first day of radiotherapy will also be acceptable. These patients will then continue to take the study drug for approximately 6 months following start of radiotherapy.
  In addition, during prophylactic phase (drug and placebo prophylactic arms) patients will have the opportunity to utilize oral 50 mg. tablets of Sildenafil Citrate in an on demand, open label, flexible dose fashion. Non-hormone patients will be offered on demand Sildenafil for approximately 12 months.
  Assessments (IIEF, IPSS, QOL) will be completed by non-hormone therapy patients at baseline (within 4 weeks of start of study treatment) and at approximately months 3, 6, 9, 12, 18 and 24 from start of radiotherapy. Testosterone assessments will take place at baseline, and months 12 and 24.
  Arms: 2

SUMMARY:
Radiation sometimes affects the ability for a person to have a normal erection. Complete loss of erections after radiation treatment can happen in 40-50% of treated patients. There are medications, like sildenafil (also known as Viagra), that can help the ability to get back erections in almost 70% of such patients.

The purpose of this study is to see if taking Viagra every day starting right before, during and for about 6 months after treatment, could reduce the risk of long-term erectile dysfunction.

DETAILED DESCRIPTION:
This protocol is a randomized prospective study comparing prophylactic and on demand Sildenafil Citrate usage administered during and after radiotherapy in combination with or without hormone therapy versus radiotherapy alone for the preservation of erectile function in potent patients with clinically localized prostate cancer. The primary objectives of this protocol are to determine if prophylactic and on demand usage of Sildenafil Citrate can preserve spontaneous erectile function as well as diminish the time to restoration of erectile function in potent men receiving radiotherapy with or without hormone therapy for localized prostate cancer. Secondary objectives of this study are: to determine whether prophylactic and on demand use of Sildenafil Citrate during therapy may improve the long-term response to the drug following treatment; to determine whether prophylactic and on demand use of Sildenafil Citrate during therapy will reduce acute and late urinary effects of radiotherapy; to determine the impact of dosimetry and radiation exposure to both the neurovascular bundle and bulb of the penis on erectile function preservation in the study population undergoing brachytherapy and hormone therapy; to asses the impact on quality of life following prophylactic and on demand Sildenafil Citrate usage in the study population; to determine the relationship between testosterone levels, erectile function and efficacy of prophylactic and on demand Sildenafil Citrate usage in the study population.

ELIGIBILITY:
Inclusion Criteria:

* To receive external beam radiation therapy and/or brachytherapy for biopsy-proven prostate cancer.
* Baseline International Index of Erectile Function (IIEF) erectile function domain score >= 17.
* Patients receiving radiotherapy with hormone therapy undergoing a maximum of 9 months of hormone therapy will be acceptable.

Exclusion Criteria:

* Baseline IIEF-EF (1-30) domain score of <17 pre-therapy
* Current routine use of erectogenic agents (use of agents > 4 times per month would constitute "routine use")
* Neoadjuvant androgen deprivation therapy started more than 1 month prior to entry into study (intake of Bicalutamide alone does not constitute exclusion from study entry)
* Have a clinically significant penile deformity in the opinion of the investigator (ie: Peyronie's Disease)
* Non-organ confined disease
* Prior prostate surgery or cryotherapy
* Prior prostate radiotherapy started more than 2 weeks prior to entry into study
* Currently taking 0.8mg Flomax daily
* Penile implant history
* Present at baseline with chronic angina requiring nitrates, angina occurring during sexual intercourse or unstable angina within the last 6 months.
* History of myocardial infarction, coronary artery bypass graft surgery or percutaneous coronary intervention within 90 days of baseline visit.
* History of significant cardiac conduction defect within 90 days of baseline visit.
* Exhibit systolic blood pressure > 170 or < 90 mm Hg or diastolic blood pressure > 100 or < 50 mm Hg at baseline visit or have a history of malignant hypertension
* Have any condition that would interfere with the subject's ability to provide informed consent or comply with study instructions, would place subject at increased risk, or might confound the interpretation of the study results
* Currently receive treatment with nitrates, cancer chemotherapy, or antiandrogens (except finasteride taken as Propecia or Proscar)
* Have a history of drug, alcohol, or substance abuse within the past 6 months, as assessed by the investigator.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2005-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Zelefsky, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Prophylactic Sildenafil Citrate With Radiotherapy: radiotherapy with hormones, questionaire assessments
  sildenafil citrate and questionaires: Hormone therapy patients will be instructed to begin the study drug simultaneously or within 1 month of start of hormone therapy. These patients will then continue to take the study drug for approximately 6 months following start of radiotherapy.In addition, during prophylactic phase (drug and placebo prophylactic arms) patients will have the opportunity to utilize oral 50 mg. tablets of Sildenafil Citrate in an on demand open label, flexible dose fashion. Hormone patients will be offered on demand Sildenafil for approximately 15-21 months.
  Hormone therapy patients will complete assessments at baseline (within 4 weeks of start of study treatment) each month (only IIEF and QOL) before start of radiotherapy, at start of radiotherapy and at months 3, 6, 9, 12 18 and 24 from start of radiotherapy. Testosterone assessments will take place at baseline, and months 12 and 24.
- Placebo With Radiotherapy: radiotherapy without hormones, questionaire assessments
  placebo tablets & questionaires: Non-hormone therapy patients will be instructed to begin the study drug 3 days prior to start of radiotherapy. Patients beginning study drug anytime between 3 days before start of radiotherapy and 2 weeks after the first day of radiotherapy will also be acceptable. These patients will then continue to take the study drug for approximately 6 months following start of radiotherapy.
  In addition, during prophylactic phase (drug and placebo prophylactic arms) patients will have the opportunity to utilize oral 50 mg. tablets of Sildenafil Citrate in an on demand, open label, flexible dose fashion. Non-hormone patients will be offered on demand Sildenafil for approximately 12 months.
  Assessments (IIEF, IPSS, QOL) will be completed by non-hormone therapy patients at baseline (within 4 weeks of start of study treatment) and at approximately months 3, 6, 9, 12, 18 and 24 from start of radiotherap
Period: Overall Study
Arm/Group | Prophylactic Sildenafil Citrate With Radiotherapy | Placebo With Radiotherapy
Started | 184 | 106
Completed | 112 | 77
Not Completed | 72 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylactic Sildenafil Citrate With Radiotherapy | Placebo With Radiotherapy | Total
Number analyzed (Participants) | 184 | 106 | 290
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 112 | 60 | 172
  >=65 years | 72 | 46 | 118
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 184 | 106 | 290
Region of Enrollment [Number; unit: participants]
  United States | 184 | 106 | 290

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Erectile Dysfunction
Description: The International Index of Erectile Function (IIEF) is used for the evaluation of male sexual function and diagnostic evaluation of Erectile Dysfunction (ED) severity. There are 5 domains of the IIEF: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. A score of 0-5 is awarded to each question of the IIEF. Total IIEF scores range from 0-75. Lower scores indicate severe erectile dysfunction (0=severe erectile dysfunction), while higher scores indicate less erectile dysfunction (75=no erectile dysfunction).
Time Frame: Baseline, 6 months, 12 months, 24 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Prophylactic Sildenafil Citrate With Radiotherapy | Placebo With Radiotherapy
Number analyzed (Participants) | 125 | 77
units on a scale
  Baseline | 64 [57.00 to 71.00] | 64 [56.75 to 69.00]
  6 mos | 59.00 [41.50 to 67.75] | 58 [35.00 to 64.00]
  12 mos | 58.00 [41.50 to 66.75] | 51 [34.50 to 63.50]
  24 months (2 years) | 58 [39.00 to 65.00] | 54.50 [29.75 to 64.75]

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Prophylactic Sildenafil Citrate With Radiotherapy | Placebo With Radiotherapy
Serious Adverse Events (participants affected / at risk) | 38/184 | 15/106
Other Adverse Events (participants affected / at risk) | 4/184 | 1/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic Sildenafil Citrate With Radiotherapy (N=184) | Placebo With Radiotherapy (N=106)
ALT, SGPT (Metabolism and nutrition disorders) | 8 (13) | 4 (7)
AST, SGOT (Metabolism and nutrition disorders) | 5 (11) | 4 (7)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (22) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (5) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Calcium, high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 12 (24) | 4 (4)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 26 (80) | 6 (7)
Hemoglobin (Blood and lymphatic system disorders) | 9 (45) | 3 (3)
INR (Blood and lymphatic system disorders) | 2 (9) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 5 (12) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PTT (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 6 (10) | 2 (2)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Sodium, high (hypernatremia) (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 3 (12) | 1 (1)
Trglycrde, high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Cholesterol,high(hypercholestremia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic Sildenafil Citrate With Radiotherapy (N=184) | Placebo With Radiotherapy (N=106)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (11) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes